CLINICAL TRIAL: NCT00045487
Title: A Phase II, Pharmacokinetic And Biologic Correlative Study of OSI-774, An EGFR Tyrosine Kinase Inhibitor, In Patients With Advanced Renal Cell Carcinoma
Brief Title: Erlotinib in Treating Patients With Advanced Kidney Cancer
Acronym: OSI-774
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000256598; IDD 01-27 (Other: University of Texas Health Science Center San Antonio); NCI-5410 (Other: National Cancer Institute (NCI))
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Results first posted 2014-01-27 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2013-12

CONDITIONS: Kidney Cancer
Keywords: recurrent renal cell cancer; stage III renal cell cancer; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OSI-774 (Experimental)
  Interventions: Drug: OSI-774

INTERVENTIONS:
Drug: OSI-774 — OSI-774 is an orally active, potent, selective inhibitor of the epidermal growth factor receptor (EGFR) tyrosine kinase.

SUMMARY:
RATIONALE: Erlotinib may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth.

PURPOSE: Phase II trial to study the effectiveness of erlotinib in treating patients who have advanced kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of erlotinib in patients with advanced renal cell carcinoma.
* Evaluate the safety and tolerability, in terms of the toxicity profile, of this drug in these patients.
* Determine the biologic activity of this drug, in terms of early disease progression, progression-free survival, 12-month survival rate, and overall survival, in these patients.
* Determine the pharmacodynamics of this drug in these patients.
* Analyze the postreceptor effects of epidermal growth factor receptor-tyrosinase kinase inhibition by this drug on cell cycle, apoptosis, and angiogenesis in tumor biopsies from these patients.
* Correlate changes in biological measurements with indices of outcome in patients treated with this drug.

OUTLINE: This is an open-label, multicenter study.

Patients receive oral erlotinib once daily on days 1-28. Courses repeat every 4 weeks for 52 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 2 months.

PROJECTED ACCRUAL: A total of 19-40 patients will be accrued for this study within 8-10 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed diagnosis of advanced renal cell carcinoma (RCC). Papillary RCC is permitted only if immunohistochemical evidence of strong (2-3+) EGFR expression.
* Disease that is recurrent or refractory to IL-2 or IFN-based therapy or new diagnosis in previously untreated patients who are not appropriate candidates to receive IL-2 -based treatment
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan.
* Prior nephrectomy or resection of metastatic lesions permitted if full surgical recovery has occurred.
* Age > 18 years Because no dosing or adverse event data are currently available on the use of OSI-774 in patients <18 years of age, children are excluded from this study but will be eligible for future pediatric single-agent trials, if applicable.
* Life expectancy of at least 12 weeks
* ECOG performance status of 0,1 or 2 or Karnofsky >60%
* Patients must have normal organ and marrow function as defined below:

Hematopoietic

1. Absolute neutrophil count at least ≥ 1,500/ul
2. Platelet ≥ 100,000/uL
3. Hemoglobin ≥ 9.0 g/dL, concomitant erythropoetin permitted Hepatic

a. Total bilirubin within normal institutional limits b. AST (SGOT)/ALT (SGPT) ≤ 2.5 times institutional upper limit of normal (≤5 times ULN if liver metastases present) Renal

a. Serum creatinine ≤ 1.5 times ULN or calculated creatinine clearance > 60 mL/min/1.73m2 Calcium

a. Corrected calcium < 12.0 mg/dl, concomitant hypocalcemic agents permitted

* Complete supportive and palliative care will continue to be provided to ameliorate signs and symptoms that were pre-existing or may arise while on study and which do not interfere with the objectives of the study. The use of erythropoietin and biphosphonates is permitted.
* Patients must have tumor blocks available for EGFR expression analysis to be eligible for treatment on this study.

Exclusion Criteria:

* History of active malignancy (other than RCC) in the past 3 years, other than nonmelanomatous skin cancer or in situ breast cancer or in situ cervical cancer.
* Patients with known brain metastases will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients may not be receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to OSI-774.
* Prior treatment with EGFR targeting therapies.
* Inability to understand the written informed consent document.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Major surgery, or significant traumatic injury occurring within 21 days prior to treatment.
* Abnormalities of the cornea based on history (e.g., dry eye syndrome, Sjogren's syndrome), congenital abnormality (e.g., Fuch's dystrophy), abnormal slit-lamp examination using a vital dye (e.g., fluorescein, Bengal Rose), and/or an abnormal corneal sensitivity test (Schirmer test or similar tear production test).
* Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease.
* Pregnant women are excluded from this study because OSI-774 is an epidermal growth factor inhibitor with the potential for teratogenic or abortifacient effects based on the data suggesting that EGFR expression is important for normal organ development. For this reason, women of childbearing potential and men must also agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with OSI-774, breastfeeding should be discontinued if the mother is treated with OSI-774.
* Because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with OSI-774. Appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated.
* Informed Consent - No study specific procedures will be performed without a written and signed informed consent document. Patients who do not demonstrate the ability to understand or the willingness to sign the written informed consent document are excluded from study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2002-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony W. Tolcher, MD, Study Chair — University of Texas Health Science Center San Antonio; Alain Mita, MD, Principal Investigator — Cedar Sinai
Locations (1):
- University of Texas Health Science Center San Antonio, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Open to accrual on 6/25/2002, closed to accrual on 4/22/2004 at The University of Texas Health Science Center at the Cancer and Therapy Research Center
Groups:
- OSI-774: OSI-774, continuous daily oral administration of 150mg until disease progression or 52 weeks duration. Dose adjustment, reduction by increments of 50mg will be made for dose-limiting toxicity.
Period: Overall Study
Arm/Group | OSI-774
Started | 41
Completed | 30
Not Completed | 11

BASELINE CHARACTERISTICS:
Groups:
- OSI-774: Once-daily oral administration for 4 weeks.
Arm/Group | OSI-774
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 32
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Ani-tumor Activity After Taking OSI-774.
Description: Antitumor activity is measured with conventional techniques such as CT, MRI or X-ray. Scans are done at baseline then evaluated for response every 2 months. All tumor measurements must be recorded millimeters (or decimal fractions of centimeters).
Time Frame: Disease progression or 52 weeks duration
Population: Intent to treat analysis.
Measure: Number; unit: participants
Arm/Group | OSI-774
Number analyzed (Participants) | 30
participants | 7 (0)

ADVERSE EVENTS:
Arm/Group | OSI-774
Serious Adverse Events (participants affected / at risk) | 4/41
Other Adverse Events (participants affected / at risk) | 0/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OSI-774 (N=41)
Skin Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Hand-Foot Syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
PT Prolongation (Cardiac disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The PI/responsible party left this institution. Additional records for completion of results entries is not available at our institution. NCI transferred the PRS record to this institution >4.5 years after the PIs left employment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No